CLINICAL TRIAL: NCT06960083
Title: A Transcranial Magnetic Stimulation Approach to Treat Misophonia
Brief Title: Transcranial Magnetic Stimulation in Misophonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Parul Jain, Fellow, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY-24-00527; 24-0489-00001 (Other Grant/Funding Number: Misophonia Research Fund)
Record Dates: First submitted 2025-04-14; First posted 2025-05-07 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Misophonia
Keywords: Misophonia; Transcranial Magnetic Stimulation; Crossover trial; Single session; EEG
MeSH Terms: conditions — misophonia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will undergo two sessions of TMS, one inhibitory and another excitatory. The immediate changes resulting from both will be measured and compared.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a TMS study. Only the technician administering TMS will be unblinded. All parties will be blinded till the end of the study. The technician is not involved in the data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inhibitory-Excitatory (IE) then Excitatory-Inhibitory (EI) (Active Comparator): Participants in this group will receive an inhibitory TMS in the first session and an excitatory TMS in the second session. The two sessions will be separated by 72 hours.
  Interventions: Other: Transcranial Magnetic Stimulation (TMS)
- Excitatory-Inhibitory (EI) then Inhibitory-Excitatory (IE) (Active Comparator): Participants in this group will receive an excitatory TMS in the first session and an inhibitory TMS in the second session. The two sessions will be separated by 72 hours.
  Interventions: Other: Transcranial Magnetic Stimulation (TMS)

INTERVENTIONS:
Other: Transcranial Magnetic Stimulation (TMS) — Transcranial Magnetic Stimulation (TMS) is an FDA-approved non-invasive brain stimulation technology. It is currently used for treating depression. Applications to other disorders such as OCD and anxiety using TMS are currently under investigation. TMS will be administered for 25 minutes.

SUMMARY:
The purpose of the project is to assess the efficacy of parietal transcranial magnetic stimulation in misophonia. N=60 participants will undergo two transcranial magnetic stimulation sessions: one inhibitory and another excitatory. During both sessions, the parietal region will be stimulated. Participants will perform computerized tasks immediately before and after the stimulation, while EEG, heart rate, and skin temperature will be recorded. These recordings will be used to assess if TMS can be used to improve tolerance to misophonia triggers.

ELIGIBILITY:
Inclusion Criteria:

* Hypersensitive to presence of a specific sound, which may be accompanied by irritation, anger/outbursts, or fear.
* Must be between the ages of 18 - 55.
* Must be fluent in English since the study's instructions, surveys, and tasks will be in English.

Exclusion Criteria:

* Axis I Psychiatric condition, past or present, as defined in DSM-V.
* Disability or medical condition that prohibits completion of study. Participants must be able to complete all study procedures to ensure optimal conditions for data analysis.
* Central Nervous System (CNS) disease, such as history of brain abnormalities (e.g., neoplasms, subarachnoid cysts), cerebrovascular disease, infectious disease (e.g., abscess), or other neurological diseases, history of head trauma (defined as loss of consciousness>3 min), or history of seizures without a resolved etiology. CNS disease and drugs that act in the peripheral or central nervous system are likely to have effects on patterns of neural activity.
* Recent or regular use of psychotropic medication (e.g., amitriptyline for migraines).
* Recent use of drugs of abuse.
* Presence of any mental implants in the head.
* Pregnant or lactating.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Unpleasantness Rating Scale | after each session, 72 hours apart (each session is 2 hours)
  Participants will be presented with a slider with extremes labelled as extremely unpleasant and extremely pleasant. Ratings will be provided for audio clips and visual cues. Full scale from 0-100, higher score indicates more unpleasantness

SECONDARY OUTCOMES:
Heart Rate | after each session, 72 hours apart (each session is 2 hours)
  The heart rate (number of beats per minute) will be measured using a wristwatch worn by the participant.
Skin Conductance Response | after each session, 72 hours apart (each session is 2 hours)
  Skin conductance, a measure capturing the amount of sweat, will be measured using a wristwatch worn by the participant.
EEG P1-N1-P2 Complex Peak Amplitude | after each session, 72 hours apart (each session is 2 hours)
  Amplitude (microvolts) of P1, N1, and P2 peaks measured in the parietal region
EEG P1-N1-P2 Complex Peak Latency | after each session, 72 hours apart (each session is 2 hours)
  Latency (milliseconds) of P1, N1, and P2 peaks measured in the parietal region
EEG Frequency Band Amplitude | after each session, 72 hours apart (each session is 2 hours)
  Amplitude (decibel) in theta (4-8 Hz), alpha (8-13 Hz), and beta (13-30 Hz) frequency bands in the parietal region
EEG Frequency Band Inter-Trial Coherence | after each session, 72 hours apart (each session is 2 hours)
  Coherence (unitless) across trials in theta (4-8 Hz), alpha (8-13 Hz), and beta (13-30 Hz) frequency bands in the parietal region

CONTACTS AND LOCATIONS:
Overall Officials: Parul Jain, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai West, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.
Access Criteria: Researchers who provide a methodologically sound proposal.
  To achieve aims in the approved proposal.
  Proposals should be directed to parul.jain@mssm.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (to be determined).